CLINICAL TRIAL: NCT01276015
Title: SPREAD AND EFFECTIVENESS OF BOTULINUM NEUROTOXIN A IN SPASTIC EQUINUS IN CEREBRAL PALSY:SHORT-TERM STUDY
Brief Title: Spread And Effectiveness Of Botulinum Neurotoxin A In Spastic Equinus In Cerebral Palsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: manager en-chief dr Caffi
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE1780
Record Dates: First submitted 2011-01-10; First posted 2011-01-13 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2009-11

CONDITIONS: Cerebral Palsy and Botulinum Toxin
Keywords: BoNT-A-botulinum neurotoxin type A; CMAP-compound muscle action potential; CP-cerebral palsy; LG-lateral gastrocnemius; MG-medial gastrocnemius; TA-tibialis anterior; PROMS-passive range of movement; MAS-modified Ashworth scale; EVGS-Edinburgh visual gait scale; GMF-CS-gross motor function classification system
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- botulinum toxin A (Experimental): botulinum toxin A diffusion in cerebral palsy
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — BoNT-A (Dysport, Ipsen) ,into the medial gastrocnemius (MG) and LG muscles unilaterally on the affected spastic hemiplegic side; dose mean± SE, 283.3± 24.7 U.. The mean dose/kg injected was 14.4± 0.8, range from 8.5 to 20 U/kg, diluted in 2.5 ml saline. frequency: once.
  Other Names: dysport, ipsen

SUMMARY:
Objectives. To study the short-term neurophysiological and clinical outcome of botulinum toxin type A(BoNT-A), injected at standard doses, and assess toxin spread to neighboring uninjected muscles in children with cerebral palsy.

Subjects and methods. The investigators studied 18 ambulatory children with dynamic equinus foot deformity (mean age 6.1 years). The gastrocnemius muscle on the affected side was injected with BoNT-A (Dysport, range from 8.9-19.4 U/kg). As the primary neurophysiological outcome measure, compound muscle action potential (CMAP) areas were assessed in the lateral gastrocnemius (LG) and tibialis anterior(TA) muscles on the treated and untreated side before BoNT-A injections (T0), and on days 10 (T10), and 30 (T30) after injections. Clinical scales were assessed and video gait was analyzed at all three time points.

Results. In all patients, CMAP areas recorded from the LG and TA muscles on the treated side decreased significantly from pre-injection values at T10 (p<0.05) and T30 (p<0.002). Assessment at both time points after injections also showed that ankle spasticity had diminished (p<0.05), equinus foot excursion increased (p<0.05), and functional gait improved (p<0.05).

Conclusion. Although BoNT-A injected at standard doses improves gait in children with spastic equinus foot the toxin spreads to uninjected leg muscles. BoNT-A treatment for cerebral palsy therefore needs individualizing according to the child's clinical features.

ELIGIBILITY:
Inclusion Criteria:

* spasticity refractory to oral medication
* patients able to walk independently or with aid
* no contraindications to BoNT-A treatment such as fixed contracture,aminoglycoside therapy and myasthenia gravis and no other neuromuscular diseases
* no orthopedic surgery before
* normal or mildly declined cognition
* previous treatment at least six months before the study

Exclusion Criteria:

* all contraindications to BoNT-A treatment

Ages: 25 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
BoNT-A injected into gastrocnemius within standard dose ranges spreads to surrounding anterior lower-limb muscles in children with CP and induces chemodenervation in injected muscles | one month
  As the primary neurophysiological outcome measure of BoNT-A induced paresis and spread, we studied changes in compound muscle action potential (CMAP) areas recorded from the lateral gastrocnemius (LG) muscle after injecting BoNT-A and from the ipsilateral tibialis anterior (TA) muscle in children with spastic hemiplegia. In line with others we considered a decreased CMAP area from LG muscle injected with BoNT-A as the neurophysiological index of BoNT-A-induced paresis

SECONDARY OUTCOMES:
the short-term clinical effect of BoNT-A injected within standard dose ranges on changes in gait in children with CP | 30 days
  As the clinical outcome measures clinical scales were assessed and video gait was analyzed before BoNT-A injections (T0), and on days 10 (T10), and 30 (T30) after injections.

CONTACTS AND LOCATIONS:
Overall Officials: laura bertolasi, md, Study Director — Universita di Verona